CLINICAL TRIAL: NCT04815434
Title: Experience and Understanding of the Mouth, Oral Health and Function Amongst
Brief Title: Experience and Understanding of the Mouth, Oral Health and Function Amongst Adults With Disabilities and Complex Health Conditions.
Acronym: FAULKS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Odontologie Clinique (CROC), Clermont-Ferrand (Unknown); Dental institute, King's College, Londres, UK (Unknown); University of Dublin, Trinity College (Other); Cork Dental School, Irlande (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 FAULKS
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-03

CONDITIONS: Adult; Disability; Chronic Disease; Oral Health
Keywords: Disable person; Chronic disease; Qualitative research; Oral Health; Sociological factors; Quality of life; Body image; Adult
MeSH Terms: conditions — Chronic Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with disabilities and complex health conditions: Interviews, experience of the mouth and oral health and function
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interviews will be conducted.

SUMMARY:
Oral health is the one of the commonest causes of health problems in the world, with almost all individuals suffering from reduced oral health at some stage over their life span. As such, oral health is a major public health issue and a major consumer of health spending. Poor oral health results in pain, infection, structural degradation, functional restrictions in chewing, swallowing and speech, change in facial appearance, social stigma, altered body image, and reduced capacity to participate in social events, amongst others. Global problems of human functioning, disability, health and environment in turn affect oral status in many complex ways (for example, ability to maintain oral hygiene, nutritional restrictions, neuromotor incapacity, dysphagia, ability to access and cooperate with treatment, etc). Disability arises from a social environment that fails to enable everyone to access it regardless of his or her impairment. Disabilities are thus socially created and not dependent on the individual's type or location of impairment. There is currently very limited qualitative research exploring perceptions of the mouth, or oral health within a social environment, from the perspective of disabled adults. No universal, holistic, comprehensive tool exists to describe oral health, the functional impact of oral health, and the environmental factors influencing oral health within the biopsychosocial model. It has been suggested that a framework for such an instrument may be supplied by the International Classification of Functioning, Disability and Health (ICF: World Health Organisation, 2001) This research seeks to address these gaps by describing perceptions of the mouth from the perspective of adults with disabilities and complex health conditions, and by linking this qualitative data to the ICF in order to assess the feasibility of using the ICF to conceptualise oral health. Adults with disabilities and complex health conditions were chosen for this ICF core set preliminary study as existing literature suggests that these respondents would accumulate not only a high level of oral health need but also experience high impact of functioning and environment on oral health.

DETAILED DESCRIPTION:
A Case Record Form will be completed during the interview with the participant and/or their carer. The form will record data relating to sociodemographics along with a subjective appreciation of general health, oral health and mental health. Sociodemographic data will include age, gender, level of education (age on completion / highest level), occupation, income band and housing tenure (own house, parent's house, institution).

An investigator will undertake the interviews. Before starting data collection, the procedure of the session will be explained and the aims of the study presented in lay terms. The investigator will state that the individual has the possibility to refuse or withdraw his/her participation at any time without consequences, and on simple request. Where possible, the interviews will take place face to face, but may be undertaken over the telephone or by video-conferencing if necessary. Audio recording will be undertaken during each interview. During the interview, field notes will be taken in order to record elements of non-verbal communication. The investigator will use a indicative topic guide covering six areas to initiate a discussion. The investigator will use a indicative topic guide covering six areas to initiate a discussion:

* How would you describe your health and your oral health?
* Do you have any health conditions which affect your mouth in any way?
* If so, which part of your mouth is affected and how?
* What is the impact of your oral health on your daily life?
* Do your living conditions or your social environment impact on your oral health in any way?
* If you had to describe the impact of your oral health on daily life to someone what would you say? Each question includes a series of prompts to assist participants in answering the question.

It is anticipated that each interview will take around 60 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years of age or over on day of data collection
* adults with self-defined disabilities and/or complex health conditions
* agreement to participate from the disabled adult or his/her carer

Exclusion Criteria:

* adults under 18 years of age
* adults without self-defined disabilities and/or complex health conditions
* refusal to participate from the disabled adult or his/her carer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with self-defined disabilities and/or complex health conditions
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Interview "experiences of the mouth in adults with disabilities and complex health conditions" | Day 1
  Interview will allow to gain understanding of the experiences of the mouth in adults with disabilities and complex health conditions
Interview "Inter-relationships between the mouth, oral health, functioning and the social environment amongst adults with disabilities and complex health conditions." | Day 1
  Interview will allow to gain understanding of the inter-relationships between the mouth, oral health, functioning and the social environment amongst adults with disabilities and complex health conditions.

SECONDARY OUTCOMES:
Interview "Ability of the ICF to contextualize experiences of oral health" | Day 1
  Interview will allow to gain insight into the ability of the ICF to contextualise experiences of oral health

CONTACTS AND LOCATIONS:
Locations (1):
- UFR d'Odontologie, Clermont-Ferrand, AURA, France

REFERENCES:
- [Derived] Bogner MS, Scambler S, Eschevins C, Faulks D. How Do Persons With Disabilities and/or Complex Health Conditions Perceive Oral Health? A Qualitative Study. Community Dent Oral Epidemiol. 2025 Feb;53(1):77-89. doi: 10.1111/cdoe.13008. Epub 2024 Oct 10. PMID 39390669